CLINICAL TRIAL: NCT00709072
Title: Relapse Following the Lidcombe Program for Preschool Children Who Stutter
Brief Title: Follow-up of Children After Stuttering Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sydney (Other)
Responsible Party: Professor Mark Onslow, The University of Sydney
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10483
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2009-06

CONDITIONS: Stuttering
Keywords: stuttering; relapse; Lidcombe Program; Preschool children
MeSH Terms: conditions — Stuttering; Recurrence | interventions — Spermine Synthase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SMS reminders
  Interventions: Behavioral: SMS (Short Message Service) reminders
- 2 (No Intervention): control group

INTERVENTIONS:
Behavioral: SMS (Short Message Service) reminders — SMS reminders sent every 2 weeks
  Arms: 1

SUMMARY:
This study aims to determine the percentage and predictors of stuttering relapse following treatment with the Lidcombe Program. It will also investigate the effectiveness of sending reminder messages to parents to assist in reducing relapse.

DETAILED DESCRIPTION:
Stuttering treatment becomes more time-consuming and less effective as children become older. Therefore it is crucial to prevent relapse following treatment in the early years. This study will investigate predictors of relapse and assess the effectiveness of a simple two-weekly user-friendly reminder to parents, about when and how to address any re-occurring stuttering after treatment. Results from the study may help to prevent stuttering relapse in this age group in the future.

ELIGIBILITY:
Inclusion Criteria:

* Completion of stage I of Lidcombe Program
* Less than 1 percent syllables stuttered at recruitment
* Means of receiving SMS email or phone reminder

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
percentage of syllables stuttered | six monthly for three years

SECONDARY OUTCOMES:
parent reported stuttering severity | six monthly for three years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Onslow, PhD, Principal Investigator — University of Sydney
Locations (1):
- Australian Stuttering Research Centre, Sydney, New South Wales, Australia